CLINICAL TRIAL: NCT04880460
Title: Effect of Magnesium Supplementation in Selective Serotonin Reuptake Inhibitors Treated Major Depressive Disorder Patients: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effect of Magnesium Supplementation in Selective Serotonin Reuptake Inhibitors Treated Major Depressive Disorder Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Sarmin Sultana, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2021/257
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2021-11

CONDITIONS: MDD
Keywords: MDD; Magnesium; DASS-21; Serum magnesium level
MeSH Terms: interventions — magnesium diglycinate

STUDY DESIGN:
Intervention Model Description: A type of intervention model describing a clinical trial in which two or more groups of participants receive different interventions. For example, a two-arm parallel assignment involves two groups of participants. One group receives drug A, and the other group receives drug B. So during the trial, participants in one group receive drug A "in parallel" to participants in the other group, who receive drug B.
Who Masked: Participant, Investigator
Masking Description: A clinical trial design strategy in which one or more parties involved in the trial, such as the investigator or participants, do not know which participants have been assigned which interventions. The type of masking was double-blind masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Active Comparator): 45 MDD patients were included in this arm who were received SSRIs and Magnesium tablets
  Interventions: Dietary Supplement: Magnesium Glycinate tablet 200mg
- Control (Placebo Comparator): 45 MDD patients were included in this arm who were received SSRIs and placebo tablets
  Interventions: Dietary Supplement: Placebo tablet 200mg

INTERVENTIONS:
Dietary Supplement: Magnesium Glycinate tablet 200mg — Magnesium glycinate tablet 200mg twice daily orally for 8 weeks along with SSRIs
  Arms: Experimental
Dietary Supplement: Placebo tablet 200mg — Placebo tablet 200mg twice daily orally for 8 weeks along with SSRIs
  Arms: Control

SUMMARY:
A randomized, double-blind, placebo-controlled trial was conducted to assess the effect of magnesium glycinate on symptoms of moderate to severe depression in 90 patients. Patients were assessed at baseline, end of the 4 weeks, and end of the 8 weeks of treatment. Patients were randomized to receive either 200 mg elemental magnesium or 200 mg placebo tablet twice daily for 8 weeks. The primary outcome measure was depression severity score assessment using Depression Anxiety Stress Scale 21 items Bangla Version (DASS-21 BV) and the secondary outcome measure was serum magnesium level estimation and side effects assessment using a preformed checklist.

DETAILED DESCRIPTION:
Major depressive disorder (MDD), is a mood disorder affecting 300 million people worldwide with a prevalence of 6.7% in Bangladesh. Depression is the main contributor to suicidal deaths and is globally ranked as the single largest contributor to non-fatal health loss. Various psychological, genetic, environmental, and biochemical factors are presumed to be involved in the causation of MDD. About 30% to 50% of patients do not respond to initial antidepressant medication, and 15% of them continue to suffer from symptoms despite the completion of multiple antidepressants and more aggressive treatment regimens, in addition to facing untoward adverse drug reactions with increasing dose. Recent trials attempted to assess the effect of magnesium in reducing depressive symptoms in MDD patients. This study evaluates whether there was any role of magnesium in reducing depressive symptoms between those who did and did not receive magnesium in 8 weeks period. Patients attending the Outpatient Department of Psychiatry, BSMMU, and diagnosed with MDD were evaluated using the DASS-21 BV for assessment of severity. Those patients who were experiencing moderate to severe symptoms (scores of 14-27) were enrolled according to inclusion and exclusion criteria. Total enrolled 90 MDD patients who have received either 200 mg elemental magnesium twice daily in the form of magnesium glycinate tablet or 200 mg placebo tablet twice daily for 8 weeks. A baseline depression severity score assessment was done using DASS-21 items and again repeated at the end of the 4 weeks and 8 weeks of treatment. Initially, baseline serum magnesium level (mg/dL) was measured and repeated again at the end of the 8 weeks of treatment. DASS-21 is a validated set of three self-report scales to measure the state of depression, anxiety, and stress, where each of the three scales contains 7 items, and each item is rated from 0 to 3. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest, anhedonia, and inertia.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed 18 years or older MDD patients of both gender according to DSM-5 at the Outpatient Department of Psychiatry, BSMMU
* Moderate to severe MDD according to DASS-21 (scores of 14-27)
* Patients prescribed only SSRIs

Exclusion Criteria:

* Patients having any other psychiatric disease, kidney disease, or gastrointestinal disease
* Taking dietary supplements in the last two months
* Taking fluoroquinolones, aminoglycosides, tetracyclines, calcium channel blockers, bisphosphonates, and skeletal muscle relaxants
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
Depression severity score assessment | 8 weeks
  Assessed the severity score of depressive symptoms using DASS-21 at baseline, end of the 4 weeks, and end of the 8 weeks treatment.
  Compared the score between before and after treatment. Compared the score between two arms. DASS21 score range from 0-28+ with the following scores: 0-9 Normal, 10-13 Mild, 14-20 Moderate, 21-27 Severe, 28+ Extremely severe.

SECONDARY OUTCOMES:
Biochemical assessment | 8 weeks
  Serum magnesium level (mg/dL) was measured at baseline and end of the 8 weeks treatment.
  Compared the serum magnesium level (mg/dL) between before and after treatment. Compare the serum magnesium level (mg/dL) between two arms.
Side effects assessment | 8 weeks
  Participants were asked about the side effects using a preformed checklist. And compare the effects between two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Md. Sayedur Rahman, MBBS, MPhil, FCPS, Study Chair — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Basic Science and Paraclinical Science of BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No